CLINICAL TRIAL: NCT01389024
Title: Hydroxyurea to Prevent Central Nervous System (CNS) Complications of Sickle Cell Disease in Children
Brief Title: Hydroxyurea to Prevent Brain Injury in Sickle Cell Disease
Acronym: HUPrevent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Washington University School of Medicine (Other); Vanderbilt University School of Medicine (Other); University of Alabama at Birmingham (Other); Children's Hospital of Philadelphia (Other); Medical University of South Carolina (Other); RTI International (Other); Columbia University (Other); Children's Mercy Hospital Kansas City (Other); Sinai Hospital of Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA_00041623; 3UL1RR025005 (NIH)
Record Dates: First submitted 2011-06-30; First posted 2011-07-07 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Stroke
Keywords: sickle cell disease; stroke; silent cerebral infarct; children
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Hydroxyurea; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxyurea (Experimental): Treatment with hydroxyurea 20 mg/kg/day increased by 5 mg/kg every 8 weeks to maximum of 35 mg/kg/day or hematologic toxicity or Absolute Neutrophil Count (ANC) <4000
  Interventions: Drug: Hydroxyurea
- Placebo (Placebo Comparator): Sucrose placebo 0.2 ml/kg/day increased to max of 0.35 ml/kg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea solution 100 mg/ml with a starting dose of 20 mg/kg/day by mouth once daily and escalation by 5 mg/kg/day every 8 weeks until hematological toxicity, an Absolute Neutrophil Count of 2000 to 4000/ul, or a maximum dose of 35 mg/kg/day.
  Other Names: Droxia; Hydrea
  Arms: Hydroxyurea
Drug: Placebo — Sucrose solution 0.2 ml/kg/day by mouth once a day with blinded dose escalation of 0.05 ml/kg/day to match the frequency of dose escalation in the hydroxyurea arm.
  Other Names: Sugar
  Arms: Placebo

SUMMARY:
This is a pilot study of hydroxyurea versus placebo to reduce central nervous system complications (abnormally fast blood flow to the brain, silent cerebral infarct or stroke) in young children with sickle cell disease. The investigators plan to identify children 12 to 48 months old without central nervous system complications and randomly assign 20 to treatment with hydroxyurea and 20 to treatment with placebo for 36 months. Neither the study doctors nor the participants will know which treatment they are receiving.

DETAILED DESCRIPTION:
Stroke, silent cerebral infarct (SCI), and cognitive impairment are frequent and highly morbid complications of sickle cell disease (SCD) in children. Current approaches to the prevention and treatment of neurological complications in SCD include screening by transcranial Doppler ultrasound (TCD) to identify children with elevated cerebral blood flow velocity who are at increased risk for strokes; these children are then typically treated with chronic transfusions indefinitely. Hydroxyurea (HU) may have beneficial effects on central nervous system (CNS) complications in SCD and reduces the frequency of painful crisis, acute chest syndrome and transfusion. The safety of HU in infants and children has been suggested in a National Institutes of Health (NIH) sponsored phase III trial; however, the exact indications for the use of HU in children remain unclear, as well as its efficacy in preventing central nervous system (CNS) complications of SCD. Our preliminary data suggest that, if the cumulative frequency of abnormal TCD, SCI and stroke could be reduced by 50%, the majority of pediatric hematologists would prescribe HU to all young children with SCD. The long term goal of this project is to perform a primary prevention trial to demonstrate the neuroprotective effect of HU and broaden the indications for HU in children. The goals of this proposal are to: 1) conduct an internal pilot randomized placebo-controlled trial of HU to reduce the CNS complications of SCD (the term internal pilot is used, as the results from the participants in the pilot will be analyzed as part of a definitive phase III trial to follow); 2) demonstrate the safety of hydroxyurea and study procedures in young children with SCD; and 3) create the leadership, network of clinical centers and other procedures necessary to conduct a definitive phase III trial demonstrating the efficacy of HU for primary prevention of the neurological complications of SCD.

The primary endpoint for the internal pilot and definitive phase III trials will be the development of abnormal TCD, SCI, transient ischemic attack (TIA) or stroke. To begin the internal pilot trial, the investigators obtained Clinical and Translational Science Award (CTSA) support at Johns Hopkins and Washington University; these sites will screen 40 participants 9-48 months of age and randomly assign and follow 20 participants for three years. Four additional centers (Children's Hospital of Philadelphia, Vanderbilt University, Children's Hospital Medical Center, Cincinnati and the University of Alabama, Birmingham) began enrollment (up to 20 patients screened and 10 participants randomly assigned per site), to provide a total of 80 participants screened, 40 randomly assigned, and a minimum of 70 participant years of follow-up. Additional sites have been added. Participants must have TCD measurements that are well below transfusion thresholds and magnetic resonance imaging (MRI) of the brain without evidence of SCI. Participants in the internal pilot will continue into a phase III trial, to complete 3 years on HU or placebo. The information from the internal pilot trial will be used to improve the design of the definitive phase III trial. The results of these studies could lead to true primary prevention of CNS complications of SCD, including abnormal TCD, SCI, neurocognitive impairment and stroke. In doing so, this study could also reduce the burden of chronic transfusions and change clinical practice by broadening the indications for HU.

ELIGIBILITY:
Inclusion Criteria for Screening

1. Participant must have sickle cell anemia (hemoglobin SS) or sickle Beta-zero (null) thalassemia (hemoglobin S-B0) as confirmed at the local institution by hemoglobin analysis after six months of age.
2. Participant must be 9 to 48 months of age. All screening procedures except MRI can be completed between 9 and 12 months of age, with the exception of the MRI, for which the child must have reached the age of 12 months.
3. Informed consent must be signed by the participant's legally authorized guardian acknowledging written consent to join the study.

Exclusion Criteria for Screening

1. History of a focal neurologic event lasting more than 24 hours with medical documentation or a history of prior overt stroke.
2. Other neurological problems, such as neurofibromatosis, lead poisoning, non-febrile seizure disorder, or tuberous sclerosis.
3. Known human immunodeficiency virus (HIV) infection.
4. Treatment with anti-sickling drugs or hydroxyurea within 3 months or anticipated treatment during the course of the study.
5. Chronic blood transfusion therapy, ongoing or planned.
6. Poor adherence likely per his/her hematologist and study coordinator based on previous compliance in clinic appointments and following advice.
7. Presence or planned permanent (or semi-permanent) metallic structures attached to their body. (e.g., braces on teeth), which their physicians believe will interfere with the MRI of the brain.
8. History of two or more TCD studies with a velocity ≥ 200 cm/sec by the non-imaging technique, or ≥185 cm/sec for the imaging technique or a indeterminate TCD.
9. Significant cytopenias [absolute neutrophil count (ANC) <1500/ul, platelets <150,000/ul, reticulocytes <80,000/ul, unless the hemoglobin is > 9 g/dl]. Cytopenias will be considered transient exclusions.
10. Other significant organ system dysfunction
11. Known allergy or intolerance of hydroxyurea
12. Significant prematurity (gestational age of < 32 weeks)

Inclusion Criteria for MRI of the Brain with Sedation

1. The parents or guardians must provide consent for sedation.

Exclusion Criteria for MRI of the Brain with Sedation

1. Failure to pass MRI screening checklist
2. Obstructive sleep apnea (OSA) and receiving therapy [e.g. continuous positive airway pressure], or being evaluated or followed by a specialist for management of severe OSA
3. Less than 12 months of age.
4. Allergic reactions such as urticaria or bronchospasm or previous adverse reactions to propofol, eggs, or soy products, if used at the participating center.
5. Allergy or previous adverse reaction to pentobarbital, if used at the participating center
6. Known major chromosomal abnormalities
7. Known airway abnormalities that would increase the risk of sedation/anesthesia.

   Temporary Exclusions
8. Room air oxygen saturation greater than or equal to 5% below the participant's baseline on the day of the MRI with sedation.
9. Room air oxygen saturation <90% on the day of the MRI with sedation.
10. Hemoglobin <6.5 g/dl (must be measured within 30 days of MRI).
11. Temperature >38˚ C on the day of sedation

8. Upper or lower respiratory infection, active bronchospasm, acute chest syndrome, splenic sequestration or other acute complications of sickle cell disease other than pain in the last 4 weeks (from resolution of symptoms) 9. Pain crisis within two weeks requiring treatment with opiates

Inclusion Criteria for Randomization

1. Participant must be 12 to 54 months of age
2. Participant must have successfully completed screening procedures (TCD, MRI of the brain, neurology exam, and cognitive evaluation)

Exclusion Criteria for Randomization

1. Participants whose MRI show a silent or overt cerebral infarct.
2. Participants who have a non-imaging TCD study with a velocity ≥ 185 cm/sec or a TCD that is indeterminate.
3. Participants with abnormal kidney function (creatinine > 0.8 mg/dl)
4. Significant cytopenias [absolute neutrophil count (ANC) <1500/ul, platelets <150,000/ul, reticulocytes <80,000/ul, unless the hemoglobin is > 9 g/dl]. Cytopenias will be considered transient exclusions.

Ages: 12 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-08-16 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Casella, MD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mercy Children's Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwiatkowski JL, Zimmerman RA, Pollock AN, Seto W, Smith-Whitley K, Shults J, Blackwood-Chirchir A, Ohene-Frempong K. Silent infarcts in young children with sickle cell disease. Br J Haematol. 2009 Aug;146(3):300-5. doi: 10.1111/j.1365-2141.2009.07753.x. Epub 2009 Jun 4. PMID 19500105
- [Background] Zimmerman SA, Schultz WH, Burgett S, Mortier NA, Ware RE. Hydroxyurea therapy lowers transcranial Doppler flow velocities in children with sickle cell anemia. Blood. 2007 Aug 1;110(3):1043-7. doi: 10.1182/blood-2006-11-057893. Epub 2007 Apr 11. PMID 17429008
- [Background] Strouse JJ, Cox CS, Melhem ER, Lu H, Kraut MA, Razumovsky A, Yohay K, van Zijl PC, Casella JF. Inverse correlation between cerebral blood flow measured by continuous arterial spin-labeling (CASL) MRI and neurocognitive function in children with sickle cell anemia (SCA). Blood. 2006 Jul 1;108(1):379-81. doi: 10.1182/blood-2005-10-4029. Epub 2006 Mar 14. PMID 16537809
- [Background] Casella JF, King AA, Barton B, White DA, Noetzel MJ, Ichord RN, Terrill C, Hirtz D, McKinstry RC, Strouse JJ, Howard TH, Coates TD, Minniti CP, Campbell AD, Vendt BA, Lehmann H, Debaun MR. Design of the silent cerebral infarct transfusion (SIT) trial. Pediatr Hematol Oncol. 2010 Mar;27(2):69-89. doi: 10.3109/08880010903360367. PMID 20201689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants were consented for the study. 18 were fully screened including an MRI of the brain. 12 participants were randomized to the two arms of the study.
Period: Overall Study
Arm/Group | Hydroxyurea | Placebo
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was not collected for non-randomized subjects.
Groups:
- Hydroxyurea: Treatment with hydroxyurea 20 mg/kg/day increased by 5 mg/kg every 8 weeks to maximum of 35 mg/kg/day or hematologic toxicity or ANC <4000
  Hydroxyurea: Hydroxyurea solution 100 mg/ml with a starting dose of 20 mg/kg/day by mouth once daily and escalation by 5 mg/kg/day every 8 weeks until hematological toxicity, an absolute neutrophil count of 2000 to 4000/ul, or a maximum dose of 35 mg/kg/day.
- Total: Total of all reporting groups
Arm/Group | Hydroxyurea | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Months] | 25.5 (11.6) | 19.7 (10.2) | 22.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 0 | 0 | 0
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Weight at screening [Mean (Standard Deviation); unit: kg] — Weight at screening in kilograms (kg).
  kg | 12.8 (2.2) | 12.4 (4.8) | 12.6 (3.6)
Hemoglobin Phenotype [Count of Participants; unit: Participants]
  Hb-SS | 6 | 5 | 11
  Hgb S-β0 thalassemia | 0 | 1 | 1
White blood cell count [Mean (Standard Deviation); unit: cells/mm^3] | 15,228 (3,250) | 14,442 (7,242) | 14,835 (5,368)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 7.8 (0.9) | 8.3 (1.1) | 8.1 (1.0)
Mean corpuscular volume [Mean (Standard Deviation); unit: fL] | 82.9 (5.1) | 79.2 (9.9) | 81.1 (7.7)
Mean corpuscular hemoglobin concentration [Mean (Standard Deviation); unit: g/dL] | 34.3 (1.6) | 33.6 (1.3) | 34.0 (1.5)
Reticulocyte count [Mean (Standard Deviation); unit: %] — Reticulocyte count as a percent (%).
  % | 17.7 (8.8) | 16.0 (7.2) | 16.9 (7.7)
Platelet count [Mean (Standard Deviation); unit: platelets per mm^3] | 417,333 (105,742) | 319,833 (88,087) | 368,583 (105,839)
Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 2.6 (1.2) | 2.0 (0.9) | 2.3 (1.1)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.25 (0.08) | 0.22 (0.04) | 0.24 (0.06)
Transcranial Doppler (TCD) TAMMV [Mean (Standard Deviation); unit: cm/sec] — TCD velocity is a measurement of cerebral blood flow velocity in cm/sec. The value presented is the time-averaged mean maximum velocity (TAMMV).
  cm/sec | 127.5 (23.9) | 109.8 (18.3) | 118.7 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Randomized Participants With Central Nervous System Complications
Description: A composite of abnormally elevated cerebral blood flow velocity as measured by transcranial Doppler ultrasound, silent cerebral infarct, or stroke.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 1 | 4
Statistical Analysis 1: Comparison: Hydroxyurea vs Placebo; Test type: Superiority; p = 0.2914, Poisson Regression; Incidence rate ratio = .216, 90% CI 2-sided [.009 to 1.66] — We calculated confidence intervals from exact Poisson regression

2. Secondary Outcome: Severe Adverse Events (SAE) Attributed to Study Procedures
Description: Number of MRIs resulting in serious adverse events. Participants can have multiple MRIs performed.
Time Frame: 3 years
Population: 18 participants underwent MRIs as part of screening. A total of 41 MRIs were performed including screening, annual or "for cause" MRIs. For this analysis, the overall number of participants analyzed is the total number of MRIs (41) performed. This outcome was not pre-specified to be collected by arm nor to evaluate treatment effect.
Measure: Count of Units; unit: MRIs
Units Other Than Participants: MRIs
Groups:
- Participants Undergoing MRIs: Of the 28 consented participants, 18 underwent MRIs at screening. An additional 23 MRIs were performed during the course of the study on the 12 randomized participants. A total of 41 MRIs were performed. Of the 41, 29 MRIs were performed under sedation.
Arm/Group | Participants Undergoing MRIs
Number analyzed (Participants) | 18
Number analyzed (MRIs) | 41
MRIs | 3

3. Secondary Outcome: Severe Adverse Events (SAE) Attributed to Sedated MRIs
Description: Number of sedated MRIs resulting in serious adverse events. Participants can have multiple MRIs performed.
Time Frame: 3 years
Population: 18 participants underwent MRIs as part of screening. A total of 41 MRIs were performed including screening, annual or "for cause" MRIs. 29 of the 41 MRIs were performed with sedation. For this analysis, the overall number of participants analyzed was the total number of sedated (29) MRIs performed. The primary intent was only to look at the effects of sedated MRI. This outcome was not pre-specified to be collected by arm nor to evaluate treatment effect.
Measure: Count of Units; unit: MRIs
Units Other Than Participants: MRIs
Groups:
- MRIs With Sedation.: Of the 28 consented participants, 18 underwent MRIs at screening. An additional 23 MRIs were performed during the course of the study. A total of 41 MRIs were performed. Of the 41, 29 MRIs were performed under sedation.
Arm/Group | MRIs With Sedation.
Number analyzed (Participants) | 18
Number analyzed (MRIs) | 29
MRIs | 3

4. Secondary Outcome: Number of Participants Randomized
Description: We will evaluate the number of participants consented and fully screened that were randomized to hydroxyurea or placebo.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Participants Completing Screening Procedures: Of the 28 consented participants, 18 completed all screening procedures.
Arm/Group | Participants Completing Screening Procedures
Number analyzed (Participants) | 18
Participants | 12

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events data was collected for all 28 consented participants during screening. 12 were randomized to the two arms of the study and collection of adverse reports was continued. Adverse events for the remainder of the consented participants who were followed only during screening were reported as a separate arm (non-randomized).
Groups:
- Screen Fails: Patients who were consented and began screening, but were not randomized
Arm/Group | Hydroxyurea | Placebo | Screen Fails
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 4/16
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=6) | Placebo (N=6) | Screen Fails (N=16)
Fever (General disorders) | 4 (8) | 5 (13) | 3 (4)
Parainfluenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Left Arm Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (3) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Splenic Sequestration (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=6) | Placebo (N=6) | Screen Fails (N=16)
Otitis Media (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Emesis (Gastrointestinal disorders) | 2 (7) | 0 (0) | 0 (0)
Anorexia (General disorders) | 1 (3) | 0 (0) | 0 (0)
Decreased appetite (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 4 (8) | 2 (3) | 1 (1)
Foot Swelling and Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Head Injury (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2) | 0 (0)
Mouth Injury (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 3 (3) | 3 (3)
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Chest X-Ray with Perihilar Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (13) | 2 (8) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (11) | 2 (9) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (12) | 1 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Discharge (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Rash (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral Icterus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hand Laceration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pica (General disorders) | 0 (0) | 2 (2) | 0 (0)
Swelling in Feet (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Hair Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Scabies (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0) | 0 (0)
Anemia with Reticulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Interpretation is limited by small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT01389024/Prot_SAP_000.pdf
  • Informed Consent Form (2013-03-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT01389024/ICF_001.pdf